CLINICAL TRIAL: NCT02856087
Title: The Effect of Ultra-low-dose Naloxone on Remifentanil-induced Postoperative Hyperalgesia - A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YSjeon_naloxone
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Pain
Keywords: acute pain; postoperative; surgery
MeSH Terms: conditions — Pain; Acute Pain | interventions — Remifentanil; Naloxone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- group LR (Placebo Comparator): low dose remifentanil (1 ng/ml of Ce) with normal saline infusion
  Interventions: Drug: Low dose remifentanil; Drug: Normal Saline
- group HR (Active Comparator): High dose remifentanil infusion (4ng/ml of Ce) with normal saline infusion
  Interventions: Drug: High dose Remifentanil; Drug: Normal Saline
- group HR-N (Experimental): remifentanil infusion at 4ng/ml of Ce with naloxone infusion
  Interventions: Drug: High dose Remifentanil; Drug: Naloxone

INTERVENTIONS:
Drug: High dose Remifentanil — remifentanil infusion at 4ng/ml of Ce
  Arms: group HR; group HR-N
Drug: Naloxone — naloxone infusion
  Arms: group HR-N
Drug: Low dose remifentanil — remifentanil infusion at 1ng/ml of Ce
  Arms: group LR
Drug: Normal Saline — normal saline infusion
  Arms: group HR; group LR

SUMMARY:
High-dose remifentanil infused intraoperative ironically results in postoperative hyperalgesia. Ultra-low dose nalxone is demonstrated to prevent these opioid-induced hyperalgesia in animal model. In this clinical trial in patients undergoing general anesthesia with remifentanil, we evaluate the effects of ultra-low-dose naloxone on remifentanil-induced hyperalgesia

DETAILED DESCRIPTION:
We enrolled adult patients undergoing thyroidectomy under general anesthesia with desflurane and remifentanil. Remifentanil was administered via target-controlled infusion and anesthetic depth was maintained keeping the BIS between 40 and 60. Patients were randomized into one of three groups depending on intraoperative doses of remifentanil and naloxone: effect-site concentrations of remifentanil 1 ng/ml (control group), 4 ng/ml (remifentanil group), and 4 ng/ml combined with infusion rate 0.8 ng/kg/min of naloxone (remifentanil and naloxone group). Postoperative mechanical pain thresholds, pain intensity, and analgesic consumption were examined during 48 h of postoperative period. The primary outcome was mechanical pain threshold measured on the peri-incisional area 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo elective thyroidectomy

Exclusion Criteria:

* consent refusal, obesity, pregnancy, hx. of thyroid surgery, neurological disorders, psychiatric disorders, hx. of drug abuse or chronic use of opioids or sedative drugs, intake of any analgesic drug within 12h before surgery.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Mechanical pain thresholds | 24hr after surgery
  Mechanical pain thresholds were assessed by von Frey filaments. The patients were asked to close their eyes during the test, and an investigator made the filament pressing the skin perpendicularly against the skin until bowing and being maintained for 1.5 seconds. The filament size was started from 0.4 g and was increased to the point until the patient perceives a clear change in sensation.

SECONDARY OUTCOMES:
Mechanical pain thresholds | 48hr after surgery
pain score | verbal numerical rating scale at 24 hr after surgery
pain score | verbal numerical rating scale at 48 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koo CH, Yoon S, Kim BR, Cho YJ, Kim TK, Jeon Y, Seo JH. Intraoperative naloxone reduces remifentanil-induced postoperative hyperalgesia but not pain: a randomized controlled trial. Br J Anaesth. 2017 Dec 1;119(6):1161-1168. doi: 10.1093/bja/aex253. PMID 29029049